CLINICAL TRIAL: NCT03386851
Title: Post-Marketing Surveillance of Safety and Effectiveness of Abilify Maintena® Injections in Korean Patients With Schizophrenia or Bipolar 1 Disorder Under the "New Drug Re-Examination"
Brief Title: Abilify Maintena PMS in Schizophrenia Patients or Bipolar 1 Disorder
Status: Completed | Type: Observational
Sponsor: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 031-402-00089
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Schizophrenia; Bipolar 1 Disorder
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

SUMMARY:
This is a Post-Marketing Surveillance (PMS) of Abilify Maintena® Injections in accordance with Korean regulations on New Drug Re-examination (i.e. New Drug Re-examination Standards: Ministry of Food and Drug Safety(MFDS) Notification).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with schizophrenia or bipolar 1 disorder
* Patients who are prescribed Abilify Maintena® Injections treatment as per investigator's medical judgment
* Patients giving written authorization to use their personal and health data and starting Abilify Maintena® Injections treatment after agreement is in place and investigators provide the explanation about objective and feature of the surveillance

Exclusion Criteria:

* Patients with known hypersensitivity to Aripiprazole or any excipients of Abilify Maintena® Injections
* Elderly patients with dementia related psychosis
* Patients who have been treated with Abilify Maintena® Injections
* Patients with score 0(Not assessed) or 1(Normal, not at all ill) in the Clinical Global Impression-Severity(CGI-S)
* Patients participating in other clinical trial
* All patients who in medical judgment of the investigator would not be appropriate for inclusion criteria in the surveillance

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Schizophrenia or bipolar 1 disorder
Sampling Method: Non-Probability Sample
Enrollment: 1030 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2021-05-25 (Actual); Study Completion 2021-05-25 (Actual)

PRIMARY OUTCOMES:
The incidence rate and the number of Adverse Events (AE)/ Adverse Drug Reactions (ADR), Serious AE/ADR, Unexpected AE/ADR | until 28 days after discontinuation

SECONDARY OUTCOMES:
Mean change from baseline to last visit in Clinical Global Impression - Severity of Illness scale (CGI-S) score. | at least 12, 24 weeks interval from baseline
Clinical Global Impression - Improvement scale (CGI-I) score at the last visit | at least 12, 24 weeks interval from baseline
Mean change from baseline to last visit inPersonal and Social Performance Scale (PSP) score. | at least 12, 24 weeks interval from baseline
Overall judgement at last visit compared to baseline, judged holistically according to clinical symptoms: "Effective", "No effect", "Worsen" | at least 12, 24 weeks interval from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- St.John of God Hospital, Gwangju, South Korea